CLINICAL TRIAL: NCT01762410
Title: An Open Label Multicentric Phase 1 Study of Oral PI3K/mTOR Inhibitor P7170 in Patients With Advanced Refractory Solid Tumors.
Brief Title: Clinical Study of Oral PI3K/mTOR Inhibitor in Patients With Advanced Refractory Solid Tumors
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision not related to patient safety
Sponsor: Piramal Enterprises Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P7170/70/11
Record Dates: First submitted 2012-12-20; First posted 2013-01-07 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Advanced Refractory Solid Tumors
Keywords: Advanced refractory solid tumors
MeSH Terms: interventions — P7170 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- P7170 (Experimental): Patients will receive study drug on a daily basis until disease progression or unacceptable toxicity in sequential cohorts following accelerated titration design.
  Interventions: Drug: P7170

INTERVENTIONS:
Drug: P7170 — Patients will receive study drug on a daily basis for twenty-one days according to the dose and schedule specified for a particular cohort of therapy. This 21 day administration will define a treatment cycle. Patients may receive consecutive treatment cycles until evidence of disease progression, intolerance of therapy, death or withdrawal from the protocol as specified.

SUMMARY:
Clinical study of oral PI3K/mTOR inhibitor P7170 in patients with advanced refractory solid tumors. The primary objective is to determine the maximum tolerated dose and dose limiting toxicity of oral PI3K/mTOR inhibitor P7170 in patients with advanced refractory solid tumors

DETAILED DESCRIPTION:
An open label multicentric Phase 1 study of oral PI3K/mTOR inhibitor P7170 in patients with advanced refractory solid tumors.The study will follow an Accelerated Titration Design (ATD) with 100% dose increments until significant toxicity as described below; followed by standard dose titration with 40% dose increments. Dose and schedule (alternate dosing regimen eg. OD, BID, intermittent) will be determined by the dose escalation outlined in the protocol and considering pharmacokinetics of the study drug determined from earlier cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Patients having histologically and/or cytologically confirmed non-haematological malignancy that is metastatic or unresectable and for which standard curative/palliative treatment does not exist or is no longer effective or is not tolerated by patient.
* Patients of either sex, of all races and ethnic groups, and more than 18 years of age.
* ECOG (Eastern Cooperative Oncology Group) performance status less than 2.
* Patients with life expectancy of at least 4 months.
* Patients with measurable or evaluable disease per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1.
* Patients must have adequate organ and marrow function as defined below:
* Absolute neutrophil count more than equal to 1500/cmm
* Platelets more than equal 100,000/cmm
* Total bilirubin within normal limits of the institution.
* AST/ALT less than equal 2.5 X institutional upper limit of normal (ULN) or less than equal 5 X institutional upper limit of normal (ULN) in the presence of liver metastases
* Creatinine less than equal 1.5 X institutional upper limit of normal (ULN)
* Women of childbearing potential and men willing to agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, during the duration of study participation and for at least 4 weeks after withdrawal from the study, unless they are surgically sterilised.
* Ability to understand and the willingness to provide a written informed consent document.

Exclusion Criteria:

1. Patients who have received any prior chemotherapy, radiotherapy, biologic/targeted anti-cancer therapy or surgery within 4 weeks (3 months for monoclonal antibodies, radioactive monoclonal antibodies or any radio- or toxin- immunoconjugates) before study drug administration and have not recovered (to < Grade 1) from the toxic effects from any prior therapy.
2. Patients having received any other investigational agents within 4 weeks prior to the date of enrolment and have not recovered completely (to < Grade 1) from the side effects of the earlier investigational agent.
3. Patients with known brain metastases (except for patients who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for two months prior to first dose of study drug.)
4. Patients with a history of myocardial infarction or uncontrolled cardiac dysfunction during the previous 6 months.
5. Patients with diabetes mellitus requiring insulin therapy at screening or patients with clinically significant diabetic complications, such as neuropathy, retinopathy, peripheral vascular disease or nephropathy.
6. Clinically significant medical condition of malabsorption, inflammatory bowel disease, or chronic diarrheal condition that might affect the absorption of the investigational agent.
7. Patients on chronic anticoagulation treatment. Prophylactic anticoagulation with low-molecular heparin is allowed.
8. Patients with inter-current illness including, but not limited to ongoing or clinically significant active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
9. Patients with a known history of allergic reaction to any other medication considered to be clinically significant by the investigator.
10. Women who are pregnant or nursing.
11. Patients with immune deficiency and at increased risk of lethal infections, for example, known h/o HIV, HBV or HCV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-11 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | End of Cycle 1 (i.e. 21 Days)
  Patients will receive study drug on a daily basis for twenty-one days according to the dose and schedule specified for a particular cohort of therapy. Toxicities observed in Cycle 1 will be considered for dose limiting toxicity (DLT) and Maximum tolerated dose (MTD)determination.

SECONDARY OUTCOMES:
Number of subject with adverse events | Until disease progression or unacceptable toxicity (expected to be 4-6 months)
  The toxic effects of the drug would be assessed from adverse events, vital signs and by clinically significant changes in the laboratory evaluations.
Pharmacokinetic profile(Cmax,Tmax and AUC) | Until disease progression or unacceptable toxicity (expected to be 4-6 months)
  The effect of dose for AUC0-t, AUC0-inf and Cmax. Tmax and T1/2 will be given as patient-wise narratives at each dose level.
Activity of P7170 based on selected biomarkers | Until disease progression or unacceptable toxicity (expected to be 4-6 months)
  Plasma samples will be used for analysis of exploratory biomarkers that are found in plasma and levels of which are likely to change in response to P7170 administration
Objective response | Until disease progression or unacceptable toxicity (expected to be 4-6 months)
  Evaluation of Response: Clinical responses will be presented patient wise for different dose levels.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony El-Khoueiry, MD, Principal Investigator — University of Southern California
Locations (4):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States
- India (3):
  - Medanta Duke Research Institute (MDRI), Gurgaon, Haryana
  - Central India Cancer Research Institute, Nagpur, Maharashtra
  - Meenakshi Mission Hospital & Research Centre, Madurai, Tamil Nadu